CLINICAL TRIAL: NCT02940236
Title: Gastric Volumes After Oral Multimodal Analgesia in the Pre-operative Setting
Brief Title: Gastric Volumes After Oral Multimodal Analgesia in the Pre-operative Setting: A Prospective Case Series
Status: Withdrawn | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elird Bojaxhi, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 16-002313
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: General Surgery
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multimodal analgesia: Patients scheduled for general surgery and requiring multimodal analgesia in preoperative period.
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Before and after patient receives oral multimodal analgesia as per standard of care, two ultrasound scans will be performed (10 minutes apart for each time element).

SUMMARY:
To assess possible risk of aspiration with pre-operative oral medications taken with "sips" of water (100ml).

ELIGIBILITY:
Inclusion Criteria:

* Patients able to take prescribed oral multimodal analgesia as per standard of care

Exclusion Criteria:

* BMI > 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients scheduled for undergo surgical procedure
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Oral multimodal analgesia and gastric volume | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No